CLINICAL TRIAL: NCT01128543
Title: A Multicenter, Open-Label, Phase II Study of Lapatinib in Combination With Vinorelbine in Subjects With ErbB2 Amplified Recurrent and Metastatic Breast Cancer
Brief Title: Lapatinib in Combination With Vinorelbine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112564
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-11

CONDITIONS: Cancer
Keywords: lapatinib; breast cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Lapatinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lapatinib 1250mg (Active Comparator): Patients will receive 1250mg lapatinib once a day for 24 weeks.
  Interventions: Drug: lapatinib and Vinorelbine
- Vinorelbine 25mg/sqm (Active Comparator): Patients will receive vinorelbine 25mg/sqm IV Day 1 and Day 8, every 3 week for 24 weeks.
  Interventions: Drug: lapatinib and Vinorelbine

INTERVENTIONS:
Drug: lapatinib and Vinorelbine — Patients will receive 1250mg lapatinib once a day and vinorelbine 25mg/sqm IV Day 1and Day 8, every 3 week for 24 weeks.

SUMMARY:
This is a Multicenter, Open-Label, Phase II Study of lapatinib in Combination with Vinorelbine in women with documented evidence of HER2/neu positive breast cancer which is metastatic or recurrent and with or without prior chemotherapy or anti-HER2/neu targeted therapy in the metastatic and relaps setting.

DETAILED DESCRIPTION:
This is a Multicenter, Open-Label, Phase II Study of lapatinib in Combination with Vinorelbine in women with documented evidence of HER2/neu positive breast cancer which is metastatic or recurrent and with or without prior chemotherapy or anti-HER2/neu targeted therapy in the metastatic and relaps setting.

Patients will receive 1250mg lapatinib once a day and vinorelbine 25mg/sqm IV Day 1and Day 8, every 3 week for 24 weeks. The study treatment will continue until patients experience disease progression or unacceptable toxicity. The primary objective of the study is the objective response rate (ORR, defined as CR + PR) and toxicity. Secondary objectives include DFS, duration of response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast.
* Patients must be > 18 years of age
* Metastatic breast cancer (stage IV) at primary diagnosis or at relapse after curative intent therapy.
* Laboratory confirmed HER2/neu overexpressing and/or amplified disease in the invasive component of the primary or metastatic lesion
* Patients must have evidence of metastatic disease, but measurable disease is not mandatory.
* The patients may have received or not prior treatment with chemotherapeutic agents including taxanes, trastuzumab or anthracycline in the adjuvant or metastatic setting is permitted.
* Prior treatments with radiation therapy in the adjuvant and/or metastatic setting are permitted provided that at least 4 weeks have elapsed since the last fraction of radiation therapy and all treatment related adverse events are < grade 1 at the time of enrollment.
* Prior radiation to a solitary metastatic lesion is permitted provided that progression post radiation has been documented.
* Patients must have life expectancy > 3 months.
* ECOG performance status 0, 1 or 2 (see Appendix II).
* Patients must have normal organ and marrow function measured within 14 days prior to enrollment as defined Table 1.
* Left ventricular ejection fraction > 50% as demonstrated by MUGA scan/echocardiogram within 4 weeks prior to enrollment.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to enrollment and must use an acceptable method of contraception for the duration of the study.

Female patients who are lactating should discontinue nursing prior to the first dose of investigational product and should refrain from nursing throughout the treatment period and for 14 days following the last dose of investigational product.

* The patient must sign the consent form prior to enrollment.
* Patients must be accessible for treatment and follow-up.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated DCIS, adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours (non-breast) curatively treated with no evidence of disease for > 5 years.
* Patients receiving ongoing anticancer treatment or other investigational anti-cancer agents for breast cancer or patients who have used an investigational drug within 30 days or 5 half-lives (if known), whichever is longer, preceding the date of enrollment.
* Patients with symptomatic CNS metastases (including leptomeningeal involvement).
* Patients with only bone metastasis.
* Patients with serious cardiac illness or condition including, but not limited to:

history of documented congestive heart failure (CHF) or systolic dysfunction (LVEF<50%) high risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV-block, supraventricular arrhythmias which are not adequately rate-controlled) unstable angina pectoris requiring anti-anginal medication clinically significant valvular heart disease evidence of transmural infarction on ECG inadequately controlled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg).

New York Heart Association (NYHA) Class III or IV functional status (see Appendix X)

* Patients who have received vinorelbine as a prior therapy in the metastatic and recurrent setting.
* Patients with serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:
* History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements.
* Active uncontrolled infection. Serious or non-healing wound, ulcer, or bone fracture.
* Patients with GI tract disease resulting in an inability to take oral medication such as but not limited to malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption (for example resection of stomach or small bowel) or uncontrolled inflammatory GI disease (e.g. Crohn's, ulcerative colitis).
* Patients receiving CYP3A4 inhibitors or inducers are not eligible unless it has been > 7 and > 14 days, respectively since the last dose of medication before the start of protocol treatment (see Appendix IX). For amiodarone in particular, dosing is prohibited for at least 6 months prior to the start of protocol treatment.
* Patients with history of allergic or hypersensitivity reactions to any study drug or their excipients or with a history of allergic reactions attributed to compounds with similar chemical composition to any of the study drugs.
* Pregnant or lactation women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Turkey (Türkiye) (5):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Diskapi / Ankara
  - GSK Investigational Site, Diyarbakır
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Kayseri

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib 1250 mg and Vinorelbine 20 mg/m^2: Participants received 1250 milligram (mg) tablets lapatinib once a day and vinorelbine 20 mg/meters squared (m^2) intravenously on Day 1 and Day 8, and every 3 weeks.
Period: Overall Study
Arm/Group | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2
Started | 29
Completed | 25
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2
Number analyzed (Participants) | 29
Age Continuous [Mean (Standard Deviation); unit: Years] | 54 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Clinical Benefit (CB) at Week 12 and Week 24
Description: Par. with CB are defined as those with complete response (CR), partial response (PR), or stable disease (SD) for >=12 or 24 weeks. Per Response Evaluation Criteria In Solid Tumors (RECIST), Version 1.1, CR is defined as the disappearance of all target lesions, PR is defined as a >=30% decrease in the sum of the longest diameter (LD) of target lesions, taking as a reference the baseline sum LD, and SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as a reference the smallest sum LD since the treatment started.
Time Frame: Week 12 and Week 24
Population: All participants randomized to receive at least one dose of study drug. Of the 29 participants enrolled in the study, 25 were evaluable for analysis; 4 participants withdrew from the study.
Measure: Number; unit: participants
Arm/Group | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2
Number analyzed (Participants) | 25
participants
  Week 12, CR | 0
  Week 12, PR | 4
  Week 12, SD | 12
  Week 24, CR | 0
  Week 24, PR | 4
  Week 24, SD | 10

2. Secondary Outcome: Progression-free Survival
Description: Per RECIST, Version 1.1, Progressive Disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From the start of treatment until disease progression, death, or discontinuation from the study (average of 102.7 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2
Number analyzed (Participants) | 25
months | 87.7 (8.7)

3. Secondary Outcome: Duration of Response
Description: Duration of response was measured in participants who experienced either a complete response or a partial response. Per RECIST, Version 1.1, complete response is defined as the disappearance of all target lesions, and partial response is defined as a >=30% decrease in the sum of the longest diameter of target lesions, taking as a reference the baseline sum longest diameter.
Time Frame: From the start of treatment until a complete response or partial response was reached (up to Week 90; average of 21.3 weeks)
Population: All participants randomized to receive at least one dose of study drug. Only those participants with a complete or partial response were evaluated.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2
Number analyzed (Participants) | 19
months | 4.6 [4.0 to 8.0]

ADVERSE EVENTS:
Arm/Group | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2 (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Candida sepsis (Infections and infestations) | 1
Urinary infection (Renal and urinary disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Lymphangitis (Blood and lymphatic system disorders) | 1
Motor deficit (Nervous system disorders) | 1
Abdominal epigastric pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1250 mg and Vinorelbine 20 mg/m^2 (N=29)
Neutropenia (Blood and lymphatic system disorders) | 18
Leucopenia (Blood and lymphatic system disorders) | 16
Diarrhea (Gastrointestinal disorders) | 14
Loss of appetite (General disorders) | 14
Anemia (Blood and lymphatic system disorders) | 11
Vomiting (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 11
High alanine transaminase (Investigations) | 9
High aspartate transaminase (Investigations) | 9
Mucositis (Respiratory, thoracic and mediastinal disorders) | 9
Eruption (Skin and subcutaneous tissue disorders) | 7
Pain (Musculoskeletal and connective tissue disorders) | 6
Constipation (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 4
Change in taste (Nervous system disorders) | 4
High alkaline phosphatase (Investigations) | 3
Fever (General disorders) | 3
Skin toxicity (Skin and subcutaneous tissue disorders) | 3
Reaction on injection region (General disorders) | 3
Hepatotoxicity (Hepatobiliary disorders) | 3
Urinary system infection (Infections and infestations) | 3
Stomatitis (Gastrointestinal disorders) | 2
Allergy (Immune system disorders) | 2
Headache (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Hand-foot syndrome (Nervous system disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Granulocytopenia (Blood and lymphatic system disorders) | 2
Weakness (General disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Cardiac toxicity (Cardiac disorders) | 2
Weight loss (Metabolism and nutrition disorders) | 2
High creatinine (Investigations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neuropathy (Nervous system disorders) | 2
Aphagia (Gastrointestinal disorders) | 2
Afebrile infection (Infections and infestations) | 1
Dysuria (Renal and urinary disorders) | 1
Axillary necrotic tissue infection (Infections and infestations) | 1
Anal fistula (Gastrointestinal disorders) | 1
Angioneurotic edema (lymphatic) (Blood and lymphatic system disorders) | 1
Leg ambustion (Skin and subcutaneous tissue disorders) | 1
Dizziness (General disorders) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Numbness at knee (Musculoskeletal and connective tissue disorders) | 1
Extravasation changes (Blood and lymphatic system disorders) | 1
Infection (Infections and infestations) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
High gamma-glutamyl transferase (Investigations) | 1
Influenza (Infections and infestations) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Bloody diarrhea (Renal and urinary disorders) | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 1
Complicated dermal toxicity (Skin and subcutaneous tissue disorders) | 1
Conjunctivitis (Eye disorders) | 1
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1
Cramp (Musculoskeletal and connective tissue disorders) | 1
Chronic fatigue syndrome (General disorders) | 1
Ear infection (Ear and labyrinth disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Flix at lession (General disorders) | 1
Meteorism (Gastrointestinal disorders) | 1
Stomach ache (Gastrointestinal disorders) | 1
Sensorial motor neuropathy (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Oral aphtha (Gastrointestinal disorders) | 1
Autonomous motor neuropathy (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Common cold (Infections and infestations) | 1
Left axillary necrotic fm tissue excision (Blood and lymphatic system disorders) | 1
Subdavien venous port implantation (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Vertigo (Nervous system disorders) | 1
Zoster (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.